CLINICAL TRIAL: NCT06890598
Title: A Phase 3, Multicenter, Double-Blind, Placebo-controlled Study Assessing the Efficacy and Safety of Olomorasib in Combination With Standard of Care Immunotherapy in Participants With Resected or Unresectable KRAS G12C-Mutant, Non-Small Cell Lung Cancer - SUNRAY-02
Brief Title: Study of Olomorasib (LY3537982) in Combination With Standard of Care in Participants With Resected or Unresectable KRAS G12C-mutant Non-Small Cell Lung Cancer
Acronym: SUNRAY-02
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18763; 2024-512302-25-00 (EU CTIS Number); J3M-MC-JZQH (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; durvalumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both Part A and B are randomized, double-blind, placebo-controlled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Olomorasib + Pembrolizumab (Experimental): Participants will receive olomorasib administered orally in combination with pembrolizumab intravenously (IV) for up to 1 year followed by olomorasib alone for up to 3 years of total treatment.
  Interventions: Drug: Olomorasib; Drug: Pembrolizumab
- Part A: Placebo + Pembrolizumab (Placebo Comparator): Participants will receive placebo administered orally in combination with pembrolizumab administered IV for up to 1 year followed by placebo alone for up to 3 years of total treatment.
  Interventions: Drug: Pembrolizumab; Drug: Placebo
- Part B: Olomorasib + Durvalumab (Experimental): Participants will receive olomorasib administered orally in combination with durvalumab administered IV for up to 1 year followed by olomorasib alone for up to 3 years of total treatment.
  Interventions: Drug: Olomorasib; Drug: Durvalumab
- Part B: Placebo + Durvalumab (Placebo Comparator): Participants will receive placebo administered orally in combination with durvalumab administered IV for up to 1 year followed by placebo alone for up to 3 years of total treatment.
  Interventions: Drug: Durvalumab; Drug: Placebo

INTERVENTIONS:
Drug: Olomorasib — Administered orally.
  Other Names: LY3537982
  Arms: Part A: Olomorasib + Pembrolizumab; Part B: Olomorasib + Durvalumab
Drug: Pembrolizumab — Administered intravenously (IV).
  Arms: Part A: Olomorasib + Pembrolizumab; Part A: Placebo + Pembrolizumab
Drug: Durvalumab — Administered IV.
  Arms: Part B: Olomorasib + Durvalumab; Part B: Placebo + Durvalumab
Drug: Placebo — Administered orally.
  Arms: Part A: Placebo + Pembrolizumab; Part B: Placebo + Durvalumab

SUMMARY:
The main purpose of this study is to assess if olomorasib in combination with pembrolizumab is more effective than the pembrolizumab and placebo combination in part A in participants with resected KRAS G12C-mutant NSCLC and to assess if olomorasib in combination with durvalumab is more effective than the durvalumab and placebo combination in part B in participants with unresectable KRAS G12C-mutant non-small cell lung cancer. The study may last up to 3 years for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of NSCLC.

  * Part A

    1. Clinical Stage II-IIIB (N2) treated with presurgical chemoimmunotherapy, with residual tumor present at time of surgery. Patients with a pathologic complete response are not eligible.
    2. Pathologic Stage II-IIIB (N2) NSCLC treated with initial upfront resection.
  * Part B - Clinical Stage III, unresectable NSCLC, without progression on concurrent platinum-based chemoradiotherapy.
* Must have disease with evidence of KRAS G12C mutation.
* Must have known programmed death-ligand 1 (PD-L1) expression
* Must have an ECOG performance status of 0 or 1.
* Able to swallow oral medication.
* Must have adequate laboratory parameters.
* Contraceptive use should be consistent with local regulations for those participating in clinical studies.
* Women of childbearing potential must

  * Have a negative pregnancy test.
  * Not be breastfeeding during treatment

Exclusion Criteria:

* Have known changes in the EGFR or ALK genes.
* Have another type of cancer that is progressing or required active treatment within the past 3 years before screening.
* Have an active autoimmune disease that required systemic treatment in the past 2 years. Endocrine replacement therapy is allowed.
* Had any immune-related side effect or allergic reaction (Grade 3 or higher) from a previous immunotherapy medicine, or any immune-related side effect greater than Grade 1 that has not resolved. This does not apply for people with hormone-related diseases who are now on stable hormone replacement therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
Part A: Disease-Free Survival (DFS) by Investigator Assessment | Randomization to disease recurrence or death from any cause (Estimated as approximately 48 months).
  DFS by Investigator Assessment
Part B: Progression-Free Survival (PFS) | Randomization to disease progression or death from any cause (Estimated as approximately 3 years).
  PFS per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by blinded independent central review (BICR)

SECONDARY OUTCOMES:
Part A & B: Overall Survival (OS) | Randomization to disease progression or death from any cause (Estimated as approximately 5 years).
  OS
Part A & B: Change from baseline in health-related quality of life (HRQoL), measured by European Organization for Research & Treatment of CancerQualityofLifeQuestionnaire-Core 30 (EORTC QLQ-C30) | Randomization through end of treatment (Estimated as approximately 3 years).
  Change from baseline in HRQoL, measured by the EORTC QLQ-C30
Part B: Objective Response Rate (ORR) per RECIST 1.1 by BICR | Randomization to disease progression or death from any cause (Estimated as approximately 3 years).
  ORR per RECIST 1.1 by BICR
Part B: Duration of Response (DOR) per RECIST 1.1 by BICR | Randomization to disease progression or death from any cause (Estimated as approximately 3 years).
  DOR per RECIST 1.1 by BICR
Part B: Disease Control Rate (DCR) per RECIST 1.1 by BICR | Randomization to disease progression or death from any cause (Estimated as approximately 3 years).
  DCR per RECIST 1.1 by BICR
Part B: Time to Response (TTR) per RECIST 1.1 by BICR | Randomization until the date that measurement criteria for CR or PR (whichever is first recorded) are first met (Estimated as approximately 3 years).
  TTR per RECIST 1.1 by BICR
Part B: Progression-Free Survival 2 (PFS2) by investigator assessment | Randomization to disease progression on next line of treatment or death from any cause (Estimated as approximately 3 years).]
  PFS2 by investigator assessment
Part B: Changes in Non-Small Cell Lung Cancer (NSCLC)-related symptoms, measured by the NSCLC-Symptom Assessment Questionnaire (SAQ) | Randomization through end of treatment (Estimated as approximately 3 years).
  Changes in NSCLC-related symptoms, measured by the NSCLC-SAQ
Part B: Time to worsening of NSCLC-related symptoms, as measured by NSCLC-SAQ | Randomization through end of treatment (Estimated as approximately 3 years).
  Time to worsening of NSCLC-related symptoms, as measured by NSCLC-SAQ
Part B: Changes in patient-reported pulmonary symptoms of cough, chest pain, and dyspnea, measured by NSCLC-SAQ | Randomization through end of treatment (Estimated as approximately 3 years).
  Changes in patient-reported pulmonary symptoms of cough, chest pain, and dyspnea, measured by NSCLC-SAQ

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (347):
- United States (74):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Infirmary Cancer Care, Mobile, Alabama
  - The University of Arizona Cancer Center - North Campus, Tucson, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - UCLA Hematology/Oncology - Santa Monica, Los Angeles, California
  - Profound Research LLC, Oceanside, California
  - University of California, Irvine (UCI) Health - UC Irvine Medical Center, Orange, California
  - Stanford Cancer Center, Palo Alto, California
  - Kaiser Permanente San Diego Mission Road, San Diego, California
  - BASS Cancer Center, Walnut Creek, California
  - Hartford Hospital (HH), Hartford, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - University of Florida - Jacksonville, Jacksonville, Florida
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Florida Cancer Specialists North, St. Petersburg, Florida
  - Comprehensive Hematology Oncology, St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialists East, West Palm Beach, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Captain James A. Lovell Federal Health Care Center, North Chicago, Illinois
  - Springfield Clinic Main Campus, Springfield, Illinois
  - Parkview Research Center at Parkview Regional Medical Center, Fort Wayne, Indiana
  - Franciscan Health, Indianapolis, Indiana
  - Baptist Health Lexington, Lexington, Kentucky
  - Baptist Health Hamburg, Lexington, Kentucky
  - CHI Saint Joseph Cancer Center - East, Lexington, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Ochsner Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - New England Cancer Specialists, Westbrook, Maine
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Reliant Medical Group, Worcester, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Jefferson Health - Cherry Hill, Cherry Hill, New Jersey
  - Sidney Kimmel Cancer Center - Washington Township, Sewell, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Northport VA Medical Center, Northport, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Interstate Medical Office Central, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University, Sidney Kimmel Cancer Center - Clinical Trials Office, Philadelphia, Pennsylvania
  - Jefferson Hospital Northeast, Philadelphia, Pennsylvania
  - AHN Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - USO - Texas Oncology - San Antonio, San Antonio, Texas
  - USO - Texas Oncology Gulf Coast, Sugar Land, Texas
  - USO - US Oncology Research Network, The Woodlands, Texas
  - The University of Vermont Medical Center Inc., Burlington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - VCU Health Adult Outpatient Pavillion, Richmond, Virginia
  - Swedish Cancer Institute - Edmonds, Edmonds, Washington
  - Swedish Medical Center, Seattle, Washington
  - Cancer Care Northwest - Vercler, Spokane Valley, Washington
  - Northwest Cancer Specialists PC, Vancouver, Washington
  - University Hospital and UW Health Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (8):
  - Icon Cancer Centre Wesley, Auchenflower
  - Sunshine Coast University Hospital, Birtinya
  - Austin Health, Heidelberg
  - ICON Cancer Centre - Kurralta Park, Kurralta Park
  - Tamworth Hospital, North Tamworth
  - Sir Charles Gairdner Hospital, Perth
  - Goulburn Valley Health, Shepparton
  - Latrobe Regional Health, Traralgon
- Austria (3):
  - Medizinische Universität Graz, Graz
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Klinik Floridsdorf, Vienna
- Belgium (4):
  - CHIREC - site delta, Auderghem
  - Antwerp University Hospital, Edegem
  - UZ Leuven, Leuven
  - AZ Delta vzw, Roeselare
- Brazil (16):
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos
  - CTO - Centro de Tratamento Oncológico, Belém
  - Oncocentro de Minas Gerais, Belo Horizonte
  - Hospital Tacchini, Bento Gonçalves
  - Centro de Pesquisa Sao Lucas, Campinas
  - Centro de Pesquisa Clínica do Instituto do Câncer do Ceará, Fortaleza
  - Hospital de Cancer de Londrina, Londrina
  - Liga Norte Riograndense Contra o Câncer, Natal
  - Hospital São Lucas da PUCRS, Porto Alegre
  - Centro de Tratamento de Tumores Botafogo para Oncoclinicas Rio de Janeiro SA, Rio de Janeiro
  - Instituto D'Or Pesquisa e Ensino, Rio de Janeiro
  - Icesp - Instituto Do Câncer Do Estado de São Paulo, São Paulo
  - Hospital Sírio Libanês, São Paulo
  - Hospital Santa Catarina - Paulista, São Paulo
  - Centro Paulista de Oncologia Clínica, São Paulo
  - Instituto D'Or de Pesquisa e Ensino (IDOR), São Paulo
- Chile (4):
  - K2 Oncology, Providencia
  - FALP, Santiago
  - Centro de Oncología de Precisión, Santiago
  - Bradfordhill, Santiago
- China (38):
  - Anyang Cancer Hospital, Anyang
  - Cancer Hospital Chinese Academy of Medical Science, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Cancer hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - Xiangya Hospital Central South University, Changsha
  - Hunan Cancer Hospital, Changsha
  - The Third People's Hospital of Chengdu (CDTPH), Chengdu
  - Sichuan Cancer hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - The Second Affiliated Hospital Chongqing Medical University, Chongqing
  - The First People's Hospital of Foshan, Foshan
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - The Second Affiliated hospital of Zhejiang University school of medicine, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jinan Central Hospital, Jinan
  - Shandong Cancer Hospital, Jinan
  - Taizhou Hospital of Zhejiang Province, Linhai
  - Liuzhou People's Hospital, Liuchow
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning
  - The Second People's Hospital of Neijiang, Neijiang
  - Shanghai Chest Hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Cancer Hospital of Shantou University Medical College, Shantou
  - ShenZhen People's Hospital, Shenzhen
  - Cancer Hospital Chinese Academy of Medical Sciences. Shenzhen Center, Shenzhen
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Tongji Hospital Tongji Medical,Science & Technology, Wuhan
  - Hubei Cancer Hospital, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Zhongshan Peoples Hospital, Zhongshan
  - ZhuZhou Central Hospital, Zhuzhou
- Czechia (2):
  - Nemocnice AGEL Ostrava - Vitkovice a.s., Ostrava
  - Fakultni nemocnice Bulovka, Prague
- France (16):
  - Hospices Civils de Lyon - Hopital Louis Pradel, Bron
  - Chu Grenoble Alpes, La Tronche
  - Centre Leon Berard, Lyon Cedex08
  - Assistance Publique Hôpitaux de Marseille - Hôpital Nord, Marseille
  - Centre Antoine-Lacassagne, Nice
  - Groupe hospitalier Paris saint Joseph, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Institut Curie, Paris
  - CHU Bordeaux Haut-Leveque, Pessac
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Hospitalier Universitaire de Rennes - Hôpital Pontchaillou, Rennes
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - CHU de Toulouse - Hopital Larrey, Toulouse
  - Hôpital Robert Schuman, Vantoux
  - Gustave Roussy, Villejuif
- Germany (20):
  - Vivantes Klinikum im Friedrichshain - Landsberger Allee, Berlin
  - Evangelische Lungenklinik Berlin, Berlin
  - Charité Campus Virchow-Klinikum, Berlin
  - DRK Kliniken Berlin Mitte, Berlin
  - Klinikum Chemnitz, Chemnitz
  - MV-Zentrum für Onkologie und Hämatologie, Cologne
  - Klinikum Köln-Merheim, Cologne
  - Onkologiezentrum Donauwörth, Donauwörth
  - HELIOS Klinikum Erfurt, Erfurt
  - Asklepios Fachkliniken München-Gauting, Gauting
  - Franziskus-Hospital Harderberg, Georgsmarienhütte
  - LungenClinic Grosshansdorf, Großhansdorf
  - Krankenhaus Martha-Maria Halle-Dölau, Halle
  - Asklepios Klinik Harburg, Hamburg
  - Thoraxklinik-Heidelberg gGmbH, Heidelberg
  - Evangelisches Krankenhaus Herne - Eickel, Herne
  - St. Elisabeth-Krankenhaus Leipzig, Leipzig
  - Klinikum Nürnberg Nord, Nuremberg
  - Robert Bosch Krankenhaus GmbH, Stuttgart
  - Universitaetsklinikum Tuebingen, Tübingen
- Greece (8):
  - Agios Savvas Regional Cancer Hospital, Athens
  - Errikos Dunant Hospital Center, Athens
  - Thoracic General Hospital of Athens "I Sotiria", Athens
  - University General Hospital of Heraklion, Heraklion
  - University General Hospital of Larissa, Larissa
  - University Hospital of Patras, Pátrai
  - Agios Loukas Clinic, Thessaloniki
  - European Interbalkan Medical Center, Thessaloniki
- Hungary (3):
  - Országos Onkológiai Intézet, Budapest
  - Budapesti Uzsoki Utcai Kórház, Budapest
  - Farkasgyepui Tudogyogyintezet, Farkasgyepű
- India (12):
  - Hemato Oncology Clinic, Ahmedabad
  - Galaxy Superspeciality Hospital, Aurangabad
  - Rajiv Gandhi Government General Hospital, Chennai
  - Sir H. N. Reliance Foundation Hospital and Research Centre, Mumbai
  - Thangam Cancer Center - Namakkal, Namakkal
  - Savera Cancer & Multi Speciality Hospital, Patna
  - Deenanath Mangeshkar Hospital & Research Centre, Pune
  - Medipoint Hospitals Pvt. Ltd., Pune
  - Malabar Cancer Centre - Thalassery, Thalassery
  - Regional Cancer Centre - Thiruvananthapuram, Thiruvananthapuram
  - Pacific Medical College & Hospital, Udaipur
  - Tata Memorial Centre - Homi Bhabha Cancer Hospital, Varanasi
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Sheba Medical Center, Ramat Gan
- Italy (10):
  - Instituto Tumori Giovanni Paolo II, Bari
  - Policlinico "G. Rodolico", Catania
  - Ospedale San Martino, Genova
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Ospedale San Gerardo-ASST Monza, Monza
  - Azienda Ospedaliera Dei Colli, Naples
  - Azienda Sanitaria Ospedaliera S Luigi Gonzaga, Orbassano
  - Istituto Nazionale Tumori Regina Elena, Rome
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Trento, Verona
- Japan (21):
  - Juntendo University Hospital, Bunkyō City
  - Tokyo Metropolitan Komagome Hospital, Bunkyō City
  - Kyushu University Hospital, Fukuoka
  - Saitama Medical University International Medical Center, Hidaka
  - Himeji Medical Center, Himeji
  - Kansai Medical University Hospital, Hirakata
  - Kanazawa University Hospital, Kanazawa
  - National Cancer Center Hospital East, Kashiwa
  - The Cancer Institute Hospital of JFCR, Kōtō City
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto
  - Shizuoka Cancer Center, Nagaizumi-cho,Sunto-gun
  - Aichi Cancer Center Hospital, Nagoya
  - Miyagi Cancer Center, Natori
  - Niigata Cancer Center Hospital, Niigata
  - Kindai University Hospital- Osakasayama Campus, Sakai
  - NHO Kinki Chuo Chest Medical Center, Sakai
  - Hokkaido University Hospital, Sapporo
  - Wakayama Medical University Hospital, Wakayama
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama
  - Kanagawa cancer center, Yokohama
  - Tottori University Hospital, Yonago
- Netherlands (7):
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek (NKI-AVL), Amsterdam
  - Amsterdam UMC, locatie VUmc, Amsterdam
  - Amphia Ziekenhuis, locatie Breda Molengracht, Breda
  - Ziekenhuis St. Jansdal, Harderwijk
  - ETZ Elisabeth, Tilburg
  - St. Antonius Ziekenhuis, locatie Utrecht, Utrecht
  - Isala, locatie Zwolle, Zwolle
- Norway (5):
  - Sorlandet Sykehus Arendal, Arendal
  - Haukeland Universitetssjukehus, Bergen
  - Drammen Sykehus, Vestre Viken HF, Drammen
  - Sykehuset Innlandet HF Gjøvik, Gjøvik
  - Oslo universitetssykehus, Radiumhospitalet, Oslo
- Poland (3):
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Kielce
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii, Poznan
  - One Day Med, Szczecin
- Portugal (4):
  - Centro Hospitalar E Universitário De Coimbra, Coimbra
  - Hospital da Luz Lisboa, Lisbon
  - Hospital CUF Porto, Porto
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE, Porto
- Romania (4):
  - Lotus-Med, Bucharest
  - SC Memorial Healthcare International SRL, Bucharest
  - Institutul Oncologic, Cluj-Napoca
  - Ovidius Clinical Hospital OCH, Ovidiu
- Slovakia (3):
  - Fakultna nemocnica s poliklinikou F.D.Roosevelta Banska Bystrica, Banská Bystrica
  - Univerzitná nemocnica Bratislava - Nemocnica Ružinov, Bratislava
  - Vychodoslovensky Onkologicky ustav a.s., Košice
- South Korea (20):
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Bupyeong-gu
  - Pusan National University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Keimyung University Dongsan Hospital, Daegu
  - Kyungpook National University Chilgok Hospital, Deagu
  - Gangnam Severance Hospital, Yonsei University Health System, Gangnam-gu
  - National Cancer Center, Goyang-si
  - Chonnam National University Hwasun Hospital, Hwasun-gun
  - Yeungnam Univeristy Medical Center, Nam-gu
  - Seoul National University Bundang Hospital, Seongnam
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University Of Korea St. Vincent's Hospital, Suwon
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (18):
  - Hospital Infanta Cristina, Badajoz
  - Parc de Salut Mar - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals, Hospitalet
  - Hospital Jerez de la Frontera, Jerez de la Frontera
  - Hospital Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - H.R.U Málaga - Hospital General, Málaga
  - Hospital Universitari Son Espases, Palma
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Clinico de Valencia, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- Sahlgrenska Universitetssjukhuset, Gothenburg, Sweden
- Switzerland (3):
  - Kantonsspital Baden, Baden
  - HFR Fribourg - Hôpital Cantonal, Fribourg
  - Kouros Moccia Oncologia, Locarno
- Taiwan (18):
  - Changhua Christian Hospital, Changhua County
  - Buddhist Dalin Tzu Chi General Hospital, Chiayi City
  - National Taiwan University Hospital Yun-Lin Branch Dou-Liou Region, Douliu
  - Hualien Tzu Chi Medical Center, Hualien City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-Da hospital, Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist
  - Far Eastern Memorial Hospital, New Taipei City
  - New Taipei Municipal TuCheng Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - Chi Mei Hospital - Liouying Branch, Tainan
  - National Taiwan University Hospital, Taipei
  - National Taiwan University Cancer Center (NTUCC), Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (11):
  - Baskent University Dr. Turgut Noyan Research and Training Center, Adana
  - Adana City Hospital, Adana
  - Sakarya University School of Medicine, Adapazarı
  - University of Health Sciences,Gulhane School of Medicine, Ankara
  - Antalya Egitim ve Arastırma Hastanesi, Antalya
  - Trakya University, Edirne
  - Gaziantep Universitesi Sahinbey Arastirma ve Uygulama Hastanesi, Gaziantep
  - İ.A.Ü VM Medical Park Florya Hastanesi, Istanbul
  - Izmir Atatürk Training and Research Hospital, Izmir
  - Marmara Universitesi Pendik Egitim Arastirma Hastanesi, Pendik
  - Samsun Medical Park Hastanesi, Samsun
- United Kingdom (7):
  - Heartlands Hospital, Birmingham
  - University Hospitals Sussex NHS Foundation Trust, East Sussex
  - Huddersfield Royal Infirmary, Huddersfield
  - Royal Marsden Hospital (Sutton), London
  - Royal Marsden Hospital (Chelsea), London
  - The Christie NHS Foundation Trust, Manchester
  - Torbay Hospital, Torquay

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Study of Olomorasib (LY3537982) in Combination With Standard of Care in Participants With Resected or Unresectable KRAS G12C-mutant Non-Small Cell Lung Cancer (SUNRAY-02) — https://trials.lilly.com/en-US/trial/585993